CLINICAL TRIAL: NCT01509378
Title: 4P Study: A Prospective Study on Predictive Quality Preferring PainFree Therapies
Brief Title: 4P Study: Predictive Quality With Painfree Therapies
Acronym: 4P
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: CH KEK-ZH-Nr. 2011-0001/4; KEK-ZH Nr 2011/0001/4 (Other: Zurich University Hospital - Switzerland)
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2016-06

CONDITIONS: Cardiac Arrhythmias
Keywords: ICD; ATP therapy; Rescue Shock therapy
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to characterize and quantify the relative effectiveness and contribution of implantable cardioverter defibrillator (ICD) therapy to the clinical outcomes under the conditions of daily practice.

Swiss, multicenter, prospective, observational study.

DETAILED DESCRIPTION:
The main role of ICD's is to stop potentially lethal ventricular tachyarrhythmias through overdrive pacing or shock, reducing the risk of sudden cardiac death. The device is programmed to detect episodes of arrhythmias, classify them according to the threat to patient, and deliver therapies to stop the arrhythmias.

The actual focus of ICD programming has been the application of fast-pacing therapies (ATP or antitachy pacing) as first therapy before applying a shock as last resort to terminate an episode. Some studies have shown the high success rate of this method in decreasing the number of shock delivered to patients. Furthermore significant improvement has been done to improve the sensitivity and specificity of the detection and discrimination algorithm.

This study will focus on the latest generation of device and their performance will be reviewed and analyzed by an Adjudication Board.

ELIGIBILITY:
Inclusion Criteria:

* Patients having an indication for a Protecta ICD or CRT-D device, or later market released ICD (first implant, replacement, or upgrade)
* Patients monitored with the Carelink monitoring system
* Patients having signed the patient informed consent form
* Patients older than 18 years

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with a life expectancy of less than 24 months
* Females, pregnant and of child bearing potential
* Patients participation to another concomitant trial
* Patients unable or not willing to provide a signed patient informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD patients primary and secondary prevention according to guidelines
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of successful and non successful therapies | 24 months follow up
  First assessment and analysis of therapy efficacy and appropriate detection and classification

SECONDARY OUTCOMES:
Number of device diagnostics alerts and device integrity alerts | 24 months follow up
  First assessment of alerts and classification
All causes hospitalizations, cardiovascular hospitalizations, death, severe adverse events (SAE) | 24 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fromer, Professor, Principal Investigator — CHUV, Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland; Mayella Favre, Study Director — Medtronic (Suisse) SA
Locations (10):
- Switzerland (10):
  - University Hospital - Basel, Basel, Canton of Basel-City
  - HFR - Hôpital Cantonal - Fribourg, Fribourg, Canton of Fribourg
  - HUG - University Hospital Geneva, Geneva, Canton of Geneva
  - Kantonsspital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - CHUV, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - GZO Spital - Wetzikon, Wetzikon, Canton of Zurich
  - Klinik Im Park - Zurich, Zurich, Canton of Zurich
  - Stadtspital TRIEMLI - Zurich, Zurich, Canton of Zurich
  - USZ - University Hospital Zurich, Zurich, Canton of Zurich
  - CardioCentro Ticino - Lugano, Lugano, Canton Ticino